CLINICAL TRIAL: NCT05212324
Title: Different Modalities in Management of Congenial Clasped Thumb
Brief Title: Management of Congenial Clasped Thumb
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Tamer Abdelkader Abdelwahed Mohammed, principal investigator, Al-Azhar University
Other Study IDs: MCCT
Record Dates: First submitted 2022-01-11; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- widening: widening of first web space by flaps, tendon transfer to extensor policis longus tendon, fractional lengthening of flexor policis longus tendon
  Interventions: Procedure: widening of first web space

INTERVENTIONS:
Procedure: widening of first web space — widening of first web space by flaps, tendon transfer to extensor policis longus tendon, fractional lengthening of flexor policis longus tendon

SUMMARY:
Congenital clasped thumb is a rare progressive flexion and adduction deformity presenting with heterogenous congenital abnormalities.(1, 2) It is confused with trigger finger deformity due to fixated flexion deformity of the thumb. In congenital trigger finger entrapment is present at A1 pulley level due to fusiform enlargement of flexor pollicis longus tendon

DETAILED DESCRIPTION:
The main problem is the deficient extensor tendon mechanism of thumb due to functional and structural causes. \

Although in congenital clasp finger deformity there are thumb flexion deformity due to extensor tendon insufficiency and muscle and skin contractions at flexor and thenar regions.

In congenital clasped thumb success of treatment depends on lesion type. Although successful results have been obtained with splinting and conservative treatment, several reconstruction methods are used due to secondarily developed contractures in neglected cases. Tendon transfers are useful in hypermobile thumb cases who have both extensor and opponents tendon deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Congenital clasped thumb
2. Cerebral palsy
3. Arthrogryposis
4. Under age of eight years old.

Exclusion Criteria:

* 1- Congenital trigger thumb. 2- Neglected adducted thumb. 3- Post traumatic extensor tendon injury. 4- Neglected congenital clasped thumb.

Ages: 2 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: when the patient diagnosed in our outpatient clinic as congenital clasped thumb we will prepare him or her to the operation after full investigation.
  surgical procedure through the skin incision designed to widen the web by flap then by do fractional lengthening of flexor policis longus tendon transfer ot extensor policis longus tendon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-02-11 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
improved hand grip degree | 3 months
  Measure the degree of thumb motion and improve function of the thumb to restore function of the hand abduction of the thumb more than 40 degree

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shreve M, Chu A. Pediatric Thumb Flexion Deformities. Bull Hosp Jt Dis (2013). 2016 Mar;74(1):97-108. PMID 26977555